CLINICAL TRIAL: NCT03233932
Title: Clinical Trial to Investigate the Safety and Pharmacokinetics/Pharmacodynamics of CKD-841 After Subcutaneous Injection in Postmenopausal Female
Brief Title: CKD-841 Pharmacokinetic/Pharmacodynamic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 155HPS14022
Record Dates: First submitted 2016-05-23; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Postmenopausal Disorder
Keywords: CKD-841; Leuplin; Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LeuplinⓡInj (Active Comparator): LeuplinⓡInj(=leuprorelin acetate 3.75mg)
  Interventions: Drug: LeuplinⓡInj
- CKD-841 (Experimental): CKD-841(=leuprorelin acetate 3.75mg)
  Interventions: Drug: CKD-841

INTERVENTIONS:
Drug: LeuplinⓡInj — Investigational drug(=LeuplinⓡInj)is prescribed single injection dose by subcutaneous to 6 of randomized subjects once.
  Arms: LeuplinⓡInj
Drug: CKD-841 — Investigational drug(=CDK-841) is prescribed single injection dose by subcutaneous to 6 of randomized subjects once.
  Arms: CKD-841

SUMMARY:
A randomized, open-label, single dose, parallel design phase I clinical trial to investigate the safety and pharmacokinetic/pharmacodynamics of CKD-841 or Leuplin Inj. 3.75mg after subcutaneous injection in postmenopausal female.

DETAILED DESCRIPTION:
To investigate the safety and pharmacokinetic/pharmacodynamics of CKD-841 or Leuplinⓡ Inj. 3.75mg after subcutaneous injection in postmenopausal female is the purpose of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy menopausal female
* β-hCG is negative at screening and before administration of investigational drug
* Infertility by sterilization operation before 5 months from screening excluding ovarian cancer, uterine cancer etc...
* Bwt ≥ 50Kg and Body Mass Index (BMI) ≥ 18.5 and < 25

Exclusion Criteria:

* History or current condition of disease related to Hepato-biliary system, renal system, nervous system, mental illness, immune system, respiratory system, endocrine system, hemato-oncology, circulatory system, musculoskeletal system or except for that, significant clinical disease
* Uncontrolled diabetes mellitus
* Pregnancy or breast feeding
* History of taking medicine such as Leuprorelin acetate or similar affiliation drug within 12 weeks before administration of investigational drug
* Has hypersensitivity to the active ingredient or excipients or same affiliation drug of the investigational drug, hypersensitivity of a medicine contained gelatin especially
* Has abnormal function of liver and kidney at screening

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Leuprorelin | From before injection to up to 1008 hours post injection
  Peak Plasma Concentration (Cmax) in ng/mL
Area Under the plasma drug Concentration-time curve to last measurement (AUClast ) of Leuprorelin | From before injection to up to 1008 hours post injection
  Area Under the plasma drug Concentration-time curve to last measurement (AUClast ) in ng•hr/mL
Area Under the plasma drug Concentration-time curve extrapolated to infinity (AUCinf) of Leuprorelin | From before injection to up to 1008 hours post injection
  Area Under the plasma drug Concentration-time curve extrapolated to infinity (AUCinf) in ng•hr/mL
Area Under the plasma drug Concentration-time curve from 7 day to last measurement (AUC7-t) of Leuprorelin | From before injection to up to 1008 hours post injection
  Area Under the plasma drug Concentration-time curve from 7 day to last measurement (AUC7-t) in ng•hr/mL
The time -to-maximal serum or plasma concentrations (Tmax) of Leuprorelin | From before injection to up to 1008 hours post injection
  The time -to-maximal serum or plasma concentrations (Tmax) in hr
Terminal half-life (t1/2) Luteinizing Hormone(LH) of Leuprorelin | From before injection to up to 1008 hours post injection
  Terminal half-life (t1/2) Luteinizing Hormone(LH) in IU/L
Follicular Stimulating Hormone(FSH) of Leuprorelin | From before injection to up to 1008 hours post injection
  Follicular Stimulating Hormone(FSH) in IU/L
Estradiol of Leuprorelin | From before injection to up to 1008 hours post injection
  Estradiol in pg/ml

SECONDARY OUTCOMES:
Safety Assessment by evaluating adverse events(AEs). | From day1 to day 56
  Assessment of the safety of subjects by evaluating adverse events(AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu 50-1, South Korea

IPD SHARING:
Plan to Share IPD: No